CLINICAL TRIAL: NCT01691391
Title: Treatment Optimization of Anti-EGFR Therapy (Cetuximab and Panitumumab) in Patients With Metastatic Colorectal Cancer Based Early 18F-FDG-PET
Brief Title: Early Biomarker With 18F-FDG PET for Treatment Optimization of Anti-EGFR Therapy in Patients With Metastatic Colorectal Cancer.
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Radboud University Medical Center (Other); Jeroen Bosch Ziekenhuis (Other); Leiden University Medical Center (Other); NKI-AvL (Unknown); Academisch Ziekenhuis Groningen (Other)
Responsible Party: Principal Investigator, C. Menke- van der Houven van Oordt, Medical Oncologist, Amsterdam UMC, location VUmc
Other Study IDs: 2010/323
Record Dates: First submitted 2012-05-15; First posted 2012-09-24 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Colorectal Cancer
Keywords: Advanced CRC
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Advanced CRC, candidates for anti-EGFR antibody monotherapy: Patients with histopathologically confirmed advanced CRC with K-Ras and BRAF wild type, aged ≥ 18 years, with a life expectancy of at least 12 weeks, who are candidates for anti-EGFR antibody monotherapy (3rd line palliative treatment).
  Interventions: Behavioral: (Early) Imaging of response with [18F-]-FDG PET-CT and kinase activity profiles

INTERVENTIONS:
Behavioral: (Early) Imaging of response with [18F-]-FDG PET-CT and kinase activity profiles — Patients will be treated with cetuximab or panitumumab. Two [18F-]-FDG PET-CT will be performed to explore early response. Patients will undergo blood sampling and two skin and tumor biopsies for kinase activity profiles.

SUMMARY:
3rd line standard treatment of patients with metastatic colorectal cancer (CRC) harboring K-ras wild type consists of anti-EGFR treatment with either cetuximab or panitumumab. This type of treatment has a modest but significant beneficial activity in this patient group with improved progression-free and overall survival. Although it is well known that patients with advanced CRC harboring a K-Ras mutation will not respond to anti-EGFR treatment, it is not understood why patients with K-Ras wild type CRC do not all benefit from this type of therapy. In order to optimize treatment of these patients as well as health care costs, it is extremely important to identify those patients who will respond to treatment with an EGFR inhibitor at an early stage.

The investigators hypothesize that the differences in response to treatment with cetuximab are due to variability in the pharmacokinetics and -dynamics of the antibody. Thus, the investigators hypothesize that patients who do not respond to anti-EGFR treatment, have insufficient drug levels in tumor tissue. The investigators hypothesize that this is due to pharmacodynamic processes such as sequestration of cetuximab in the liver which expresses high levels of EGF receptor.

The phase I part of the study was fulfilled after inclusion of 36 patients to evaluate the potential applicability of the 89Zr-cetuximab PET as predictive marker for (absence of) response to cetuximab. Along with this analysis, FDG-PET evaluation before and after 1 administration of cetuximab was being performed. While we observed no correlation of 89Zr-cetuximab tumor uptake with clinical benefit in these 36 patients, we did find a clinical significant predictive value for the absence of response with early 18F-FDG-PET with the lack of clinical benefit at 2 months of treatment in this group of patients. Early 18F-FDG PET response evaluation shows great potential to be a clinically applicable tool to stop an ineffective treatment in a very early phase after one administration of treatment. Such an early predictor is unprecedented in clinical daily practice and will 1) avoid unnecessary toxicity of inactive treatment, 2) will lead to faster prescription of a potentially active alternative treatment and 3) will reduce costs by preventing administration of inactive treatment. In order to provide solid evidence for this new approach, we aim to validate early 18F-FDG-PET as a predictive imaging strategy to identify non-responders in part 2 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Advanced colorectal adenocarcinoma
* Subjects must have been treated according to standard care with a fluoropyrimidine (e.g. fluorouracil or capecitabine), irinotecan, and oxaliplatin or had contra-indications to treatment with these drugs.
* Age ≥18 years.
* Histological or cytological documentation of cancer is required.
* Tumor material must be tested wild type for the K-Ras gene.
* Subjects have at least one measurable lesion outside the liver. Lesions must be evaluated by CT-scan or MRI according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1).
* ECOG Performance Status of 0, 1 or 2
* Adequate liver and renal functions as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:

  * Total bilirubin ≤ 1.5 times the upper limit of normal
  * ALT and AST ≤ 2.5 times upper limit of normal (≤ 5 times upper limit of normal for subjects with liver involvement of their cancer)
  * Serum creatinin ≤ 1.5 times upper limit of normal or a calculated creatinin clearance ≥ 50 ml/min
* Signed informed consent must be obtained prior to any study specific procedures.

Exclusion Criteria:

* Previous exposure to an anti-EGFR therapy
* Significant skin condition interfering with treatment
* Insulin dependency
* Pregnant or breast-feeding subjects. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. Both men and women enrolled in this trial must agree to use adequate barrier birth control measures (e.g., cervical cap, condom, and diaphragm) during the course of the trial. Oral birth control methods alone will not be considered adequate on this study, because of the potential pharmacokinetic interaction between study drug and oral contraceptives. Concomitant use of oral and barrier contraceptives is advised. Contraception is necessary for at least 6 months after receiving study drug.
* Concurrent anticancer chemotherapy, immunotherapy or investigational drug therapy during the study or within 4 weeks of the start of study drug.
* Radiotherapy to the target lesions during study or within 4 weeks of the start of study drug. Palliative radiotherapy will be allowed.
* Major surgery within 28 days of start of study drug.
* Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results.
* Any condition that is unstable or could jeopardize the safety of the subject and their compliance in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histopathologically confirmed advanced CRC with K-Ras and BRAF wild type, aged ≥ 18 years, with a life expectancy of at least 12 weeks, who are candidates for anti-EGFR antibody monotherapy (3rd line palliative treatment).
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2012-01; Primary Completion 2020-11-03 (Actual); Study Completion 2020-11-03 (Actual)

PRIMARY OUTCOMES:
The predictive value of 18F-FDG-PET for the absence of response compared to the lack of clinical benefit at convential CT at 2 months | assessed up to 2 months; date of first CT-scan evaluation
  The predictive value of 18F-FDG-PET for the absence of response compared to the lack of clinical benefit at convential CT at 2 months

SECONDARY OUTCOMES:
Grade of skin toxicity | every 4 weeks until progressive disease
  Grade of skin toxicity as measured by predefined criteria (see below).

CONTACTS AND LOCATIONS:
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] van Helden EJ, Hoekstra OS, Boellaard R, Roth C, Mulder ER, Verheul HM, Menke-van der Houven van Oordt CW. Early 18F-FDG PET/CT Evaluation Shows Heterogeneous Metabolic Responses to Anti-EGFR Therapy in Patients with Metastatic Colorectal Cancer. PLoS One. 2016 May 19;11(5):e0155178. doi: 10.1371/journal.pone.0155178. eCollection 2016. PMID 27196139